CLINICAL TRIAL: NCT00905359
Title: A Multicenter Prospective Randomized Controlled Clinical Trial to Evaluate the Effectiveness and Safety of the Aperius™ PercLID™ System Versus Standalone Decompressive Surgery in Degenerative Lumbar Spinal Stenosis With Neurogenic Intermittent Claudication
Brief Title: Neurogenic Intermittent Claudication Evaluation Study
Acronym: NICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP 0002 AP
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aperius™ PercLID™ System (Active Comparator): Aperius™ PercLID™ System arm. Patients randomized to this arm will undergo treatment with the Aperius™ PercLID™ System.
  Interventions: Procedure: Aperius™ PercLID™ System
- Standalone Decompressive Surgery (Active Comparator): Patients randomized to this arm will receive Standalone Decompressive Surgery, defined as decompressive surgery without instrumentation or fusion.
  Interventions: Procedure: Standalone Decompressive Surgery

INTERVENTIONS:
Procedure: Aperius™ PercLID™ System — Aperius™ PercLID™ System: implantation with the Interspinous Process Device Aperius.
  Arms: Aperius™ PercLID™ System
Procedure: Standalone Decompressive Surgery — Lumbar decompressive surgery without instrumentation or fusion
  Arms: Standalone Decompressive Surgery

SUMMARY:
The objective of the NICE study is to provide clinical evidence proving that the Aperius™ PercLID™ System is safe and non-inferior to standalone decompressive surgery with regards to clinical outcomes in patients suffering from Degenerative Lumbar Spinal Stenosis with Neurogenic Intermittent Claudication, relieved by flexion.

DETAILED DESCRIPTION:
The NICE study is a Multicenter Prospective Randomized Controlled Clinical Trial to Evaluate the Effectiveness and Safety of the Aperius™ PercLID™System Versus Standalone Decompressive Surgery in Degenerative Lumbar Spinal Stenosis with Neurogenic Intermittent Claudication.

DLSS patients suffering from NIC that would be candidates for surgical treatment without stabilization and/or fusion can be offered participation in the study. After randomization, patients will be treated with either the Aperius™ PercLID™ System or Standalone Decompressive Surgery (SDS). A sample size recalculation reduced the amount of patients to be enrolled from 280 to 128 in both treatment group.

The patient will undergo a study visit at screening / baseline and at 14 days, 6 weeks, 6, 12 and 24 months after surgery. Safety data will be collected during surgery and throughout the 24 months follow up. Procedural details will be collected during surgery and also duration of hospital stay will be collected. At screening / baseline and all follow up visits a physical examination will be performed, the use of pain medication will be documented and the subject will be asked to complete a pain VAS scale (back - leg - buttock / groin pain) and questionnaires (SF36 v2 and Zurich Claudication Questionnaire).

Study subjects are required to undergo X-ray, CT and MRI and fluoroscopy procedures at specified time points during the study.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptomatic DLSS
* Presence of NIC
* Patient would be candidate for Standalone Decompressive Surgery
* Patient has signed Informed Consent form (ICF)
* Patient is 21 years old or older

Exclusion Criteria:

* Previous lumbar surgery
* Patient is candidate for instrumented Decompressive Surgery
* Patient has back pain without leg pain
* Degenerative Spondylolisthesis greater than grade 1 (Meyerding)
* Symptomatic DLSS at more than 2 levels in the lumbar region
* Spinal stenosis is present at L5-S1 level

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2010-01; Primary Completion 2014-09 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Le Huec, Prof., Principal Investigator — CHU Pellegrin Tripode
Locations (19):
- Pindara Specialist Suite, Benowa, Queensland, Australia
- Belgium (5):
  - Ziekenhuis St. Jan - Orthopedie, Bruges
  - Clinique Parc Leopold - Neurochirurgie, Brussels
  - CHU Tivoli - Neurochirurgie, La Louvière
  - Clinique Saint Joseph - Neurochirurgie, Liège
  - Centre hospitalier du Grand Hornu - Orthopédie / Traumatologie, Mons
- France (3):
  - Centre Universitaire Pellegrin Tripode -Orthopédie-Traumatologie, Bordeaux
  - Hôpital Roger Salengro - Clinique de Neurochirurgie, Lille
  - CHU de Nice Hôpital Pasteur - Neurochirurgie, Nice
- Germany (2):
  - Neurochirurgische Klinik - Campus Benjamin Franklin, Berlin
  - Klinikum rechts der Isar der TU München - Neurochirurgie, München
- Landspitali - National hospital of Iceland, Reykjavik, Iceland
- Italy (2):
  - Azienda Ospedaliera Sant'Andrea - Neurochirurgia, Rome
  - Ospedale di Circolo - Ortopedia e Traumatologia, Varese
- Poland (2):
  - Municipal Hospital - Szpital Miejski, Torun
  - Szpital Kliniczny Dziecatka Jezus - Orthopaedics, Warsaw
- Singapore General Hospital - Orthopaedic Surgery, Singapore, Singapore
- Ortopedmottagningen SU/Sahlgrenska, Gothenburg, Sweden
- Woodend Hospital - Department of Orthopaedics, Aberdeen, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Aperius™ PercLID™ System: Patients randomized to this arm underwent treatment with the Aperius™ PercLID™ System.
- Standalone Decompressive Surgery: Patients randomized to this arm received Standalone Decompressive Surgery, defined as decompressive surgery without instrumentation or fusion.
Period: Overall Study
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Started | 82 | 81
12 Months Follow up | 68 | 72
24 Months Follow up | 58 | 65
Completed | 58 | 65
Not Completed | 24 | 16
Not completed — Lost to Follow-up | 17 | 10
Not completed — Death | 2 | 0
Not completed — Withdrawal consent | 5 | 6

BASELINE CHARACTERISTICS:
Population: Per statistical analysis plan, populations excluded patients who withdrew consent during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.29 (10.91) | 64.59 (10.22) | 64.94 (10.55)
Gender [Count of Participants; unit: Participants]
  Female | 41 | 37 | 78
  Male | 36 | 38 | 74
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.54 (3.50) | 28.07 (3.54) | 28.31 (3.51)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change From Baseline in Physical Function at 1 Year Follow-up Using the Patient Completed Zurich Claudication Questionnaire
Description: ZCQ is a validated outcomes instrument specific to lumbar spinal stenosis, and captures data in 3 distinct domains: Physical function (PF), Symptom Severity (SS), and post-treatment Patient Satisfaction (PS).PF score is the mean score of five physical function questions of ZCQ, ranging from 1 to 4. A lower score represents a better outcome/condition. Mean percentage change from baseline in Physical Function at 1 year follow-up was reported.
Time Frame: 1 year
Population: Per-protocol analysis (subjects who were not performed surgical procedure as assigned per randomization were excluded).
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 72 | 73
percentage change from baseline | -32.31 (32.06) | -37.48 (22.79)
Statistical Analysis 1: Comparison: Aperius™ PercLID™ System vs Standalone Decompressive Surgery; Test type: Non-Inferiority or Equivalence — t-test analysis performed using Multiple imputation and one-sided p-value testing non-inferiority of the percentage change from baseline at 10%. One-sided p-value is significant if <0.025 or the upper limit of the CI is less than 10%; p = 0.172, t-test, 1 sided

2. Secondary Outcome: Mean Percentage Change From Baseline in Physical Function, Using Patient Completed Zurich Claudication Questionnaire
Description: ZCQ is a validated outcomes instrument specific to lumbar spinal stenosis, and captures data in 3 distinct domains: Physical function (PF), Symptom Severity (SS), and post-treatment Patient Satisfaction (PS).PF score is the mean score of five physical function questions of ZCQ, ranging from 1 to 4. A lower score represents a better outcome/condition. Mean percentage change from baseline in Physical Function at 14 days, 6 weeks, 6 months, and 24 months was reported.
Time Frame: 14 days, 6 weeks, 6 months, and 24 months
Population: Per-protocol population analysis (subjects who were not performed surgical procedure as assigned per randomization were excluded).
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 72 | 73
percentage change from baseline
  at 14 days | -19.70 (28.87) | -18.52 (28.07)
  at 6 weeks | -32.17 (27.36) | -34.60 (24.19)
  at 6 months | -34.94 (25.92) | -38.11 (21.70)
  at 24 months | -37.86 (21.72) | -35.15 (22.78)

3. Secondary Outcome: Mean Percentage of Change From Baseline in Symptom Severity of the Patient Completed Zurich Claudication Questionnaire
Description: ZCQ is a validated outcomes instrument specific to lumbar spinal stenosis, and captures data in 3 distinct domains: SS, PF, and post-treatment PS. SS Score is based on seven questions (overall pain, pain frequency, pain in the back, pain in the leg, numbness, weakness, and balanced disturbance) in ZCQ. The first 6 questions are scored 1 to 5. Balance disturbance is scored in a 1-3-5 scale. The SS score is the mean of all answered items in the questionnaire, ranging from 1 to 5. A lower score represents a better outcome/condition. Mean percentage of change from baseline in Symptom Severity is reported.
Time Frame: 14days, 6 week, 6 months, 12 months, 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 72 | 73
percentage change from baseline
  At 14 days (n=67, 66) | -34.38 (19.32) | -27.92 (19.32)
  At 6 weeks (n=66, 68) | -35.72 (22.08) | -36.38 (19.26)
  at 6 months (n=60, 62) | -33.86 (21.70) | -34.18 (19.84)
  At 12 months (n=60, 63) | -31.24 (26.85) | -36.40 (24.53)
  At 24 months (n=50, 57) | -40.25 (21.91) | -32.78 (23.89)

4. Secondary Outcome: Patient Satisfaction (PS) Scores of Zurich Claudication Questionnaire
Description: PS score is the mean score of 6 questions of ZCQ, ranging from 1 to 4 if the number of responses exceeded four. A lower score represents a better outcome. Patients with PS score less than 2.5 at postoperative evaluation were considered positive, which implied that patients were satisfied with their treatment.
Time Frame: 14 days, 6 weeks, 6 months, 12 months, and 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 72 | 73
units on a scale
  PS score at 14 days | 1.76 (0.55) | 1.77 (0.59)
  PS score at 6 weeks | 1.71 (0.49) | 1.64 (0.48)
  PS score at 6 months | 1.73 (0.63) | 1.67 (0.58)
  PS score at 12 months | 1.73 (0.66) | 1.73 (0.70)
  PS score at 24 months | 1.68 (0.68) | 1.72 (0.69)

5. Secondary Outcome: Mean Percentage Change of Visual Analog Scale (VAS) From Baseline in Leg Pain
Description: Patients rated their leg pain using Visual Analog Scale (VAS) from 0 to 10, higher values represents a worse pain. Mean percentage change of VAS scores from baseline in leg pain is reported.
Time Frame: 14 days, 6 weeks, 6 months, 12 months, and 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 72 | 73
percentage of change from baseline
  at 14 days | -67.62 (35.57) | -57.64 (35.70)
  at 6 weeks | -65.14 (32.49) | -67.65 (35.54)
  at 6 months | -56.10 (37.97) | -66.75 (34.62)
  At 12 months | -59.20 (35.75) | -66.41 (31.98)
  At 24 months | -70.71 (34.44) | -66.55 (31.11)

6. Secondary Outcome: Mean Percentage Changes From Baseline in Quality of Life Using the Patient-completed SF-36 Questionnaire
Description: The SF-36 questionnaire was used to assess the quality of life. The SF-36 results were summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for PCS and MCS is between 0 and 100, with higher scores denoting better quality of life. Mean percentage changes of SF-36 PCS and MCS from baseline are reported.
Time Frame: 14 days, 6 weeks, 6 months, 12 months, and 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 72 | 73
percentage of change from baseline
  percentage change of PCS at 14 days | 35.93 (50.06) | 27.40 (38.39)
  percentage change of PCS at 6 weeks | 52.28 (50.37) | 46.16 (42.02)
  percentage change of PCS at 6 months | 53.95 (53.04) | 42.52 (39.00)
  percentage change of PCS at 12 months | 47.83 (53.69) | 44.82 (37.77)
  percentage change of PCS at 24 months | 51.53 (49.37) | 39.27 (37.17)
  percentage change of MCS at 14 days | 18.74 (31.60) | 23.42 (39.98)
  percentage change of MCS at 6 weeks | 25.27 (35.05) | 26.57 (46.69)
  percentage change of MCS at 6 months | 20.21 (40.35) | 25.90 (44.57)
  percentage change of MCS at 12 months | 18.21 (34.86) | 23.90 (40.89)
  percentage change of MCS at 24 months | 20.05 (31.80) | 21.74 (40.81)

7. Secondary Outcome: Number of Subjects Requiring Secondary Surgical Intervention
Time Frame: Overall study period, up to 24 months
Population: Safety population: All patients who were operated within this study (either by an APERIUS® procedure or by SDS).
Measure: Number; unit: participants
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 77 | 75
participants | 16 | 6

8. Secondary Outcome: Percentage of Subjects With Serious Adverse Device Effects
Time Frame: Overall study period, up to 24 months
Population: Safety population: All patients who were operated within this study (either by an APERIUS® procedure or by SDS).
Measure: Number; unit: percentage of subjects
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 77 | 75
percentage of subjects | 3.9 | 0.0

9. Secondary Outcome: Changes in Stenosis of the Spinal Canal Assessed by Magnetic Resonance Imaging (MRI) at the Follow-up Time Points
Description: The lumen sizes of the spinal central canal were reported for the changes in stenosis of the spinal canal assessed by Magnetic Resonance Imaging (MRI) at the follow-up time points.
Time Frame: baseline, 12 months, and 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 72 | 73
mm^2
  First level operated at baseline (n=61, 62) | 7.81 (3.33) | 8.20 (2.97)
  First level operated at 12 months (n=53, 56) | 9.55 (3.61) | 13.40 (5.41)
  First level operated at 24 months (n=48, 49) | 10.43 (3.54) | 13.80 (5.32)
  Second level operated at baseline (n=28, 29) | 7.30 (2.91) | 7.72 (3.10)
  Second level operated at 12 months (n=26, 25) | 9.44 (4.45) | 15.21 (5.52)
  Second level operated at 24 months (n=21, 23) | 10.20 (4.94) | 16.18 (5.36)

10. Secondary Outcome: Bony Structure Changes of Spinous Process Assessed by CT at the Follow-up Time Points
Description: Number of subjects who had abnormal bony structure of Spinous process was reported for bony structure changes of Spinous process assessed by CT at the follow-up time points.
Time Frame: baseline, 12 months, and 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 72 | 73
participants
  First level operated at baseline | 3 | 1
  First level operated at 12 months | 2 | 15
  First level operated at 24 months | 1 | 7
  Second level operated at baseline | 3 | 2
  Second level operated at 12 months | 5 | 13
  Second level operated at 24 months | 3 | 6

11. Secondary Outcome: Correlation Between Changes in Spinal Central Canal Stenosis and Changes in Patient Reported Outcomes-Back Pain
Time Frame: 12 months and 24 months
Population: Intention to treat population analysis: all randomized patients who were operated, and had at least one post-operative assessment.
Measure: Number; unit: correlation coefficient
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 77 | 75
correlation coefficient
  First operated level at 12 months (n=49, 52) | -0.222 | -0.144
  First operated level at 24 months (n=42, 39) | -0.013 | -0.229
  Second operated level at 12 months (n=25, 20) | -0.200 | 0.026
  Second operated level at 24 months (n=17, 17) | 0.029 | 0.103

12. Secondary Outcome: Correlation Between Changes in Spinal Central Canal Stenosis and Changes in Patient Reported Outcomes-leg Pain
Time Frame: 12 months and 24 months
Population: as for outcome 11
Measure: Number; unit: correlation coefficient
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 77 | 75
correlation coefficient
  First operated level at 12 months (n=49, 52) | -0.210 | -0.264
  First operated level at 24 months (n=42, 39) | 0.051 | -0.276
  Second operated level at 12 months (n=25, 20) | 0.181 | -0.050
  Second operated level at 24 months (n=17, 17) | -0.065 | -0.287

13. Secondary Outcome: Correlation Between Changes in Spinal Central Canal Stenosis and Changes in Patient Reported Outcomes-ZCQ Physical Function
Time Frame: 12 months and 24 months
Population: as for outcome 11
Measure: Number; unit: correlation coefficient
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 77 | 75
correlation coefficient
  First level operated at 12 months (n=48, 50) | -0.179 | -0.242
  First level operated at 24 months (n=41, 37) | 0.193 | -0.163
  Second operated level at 12 months (n=24, 20) | -0.016 | 0.145
  Second operated level at 24 months (n=17, 17) | 0.173 | -0.104

14. Secondary Outcome: Correlation Between Changes in Spinal Central Canal Stenosis and Changes in Patient Reported Outcomes-ZCQ Symptom Severity
Time Frame: 12 months and 24 months
Population: as for outcome 11
Measure: Number; unit: correlation coefficient
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 77 | 75
correlation coefficient
  First operated level at 12 months (n=48, 50) | -0.091 | -0.196
  First operated level at 24 months (n=40, 37) | 0.177 | -0.367
  Second operated level at 12 months (n=24, 20) | 0.114 | 0.020
  Second operated level at 24 months (n=16, 17) | -0.368 | -0.230

15. Secondary Outcome: Number of Patients With Improvement of Symptoms, Symptoms Recurrence, Decreased Therapeutic Response, no Therapeutic Response and Treatment Failure at 14 Days, 6 Weeks, 6, 12 and 24 Months
Time Frame: 14 days, 6 weeks, 6 months, 12 months, and 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Number analyzed (Participants) | 72 | 73
participants
  Improvement of symptoms at 14 days | 34 | 30
  Improvement of symptoms at 6 weeks | 46 | 49
  Improvement of symptoms at 6 months | 43 | 46
  Improvement of symptoms at 12 months | 41 | 43
  Improvement of symptoms at 24 months | 38 | 42
  Symptom recurrence at 14 days | 0 | 0
  Symptom recurrence at 6 weeks | 2 | 3
  Symptom recurrence at 6 months | 9 | 9
  Symptom recurrence at 12 months | 11 | 13
  Symptom recurrence at 24 months | 8 | 8
  Decreased therapeutic response at 14 days | 0 | 0
  Decreased therapeutic response at 6 weeks | 12 | 5
  Decreased therapeutic response at 6 months | 15 | 14
  Decreased therapeutic response at 12 months | 10 | 12
  Decreased therapeutic response at 24 months | 10 | 11
  No therapeutic response at 14 days | 0 | 0
  No therapeutic response at 6 weeks | 18 | 12
  No therapeutic response at 6 months | 9 | 7
  No therapeutic response at 12 months | 7 | 6
  No therapeutic response at 24 months | 5 | 7
  Treatment failure at 14 days | 0 | 0
  Treatment failure at 6 weeks | 0 | 0
  Treatment failure at 6 months | 0 | 0
  Treatment failure at 12 months | 0 | 1
  Treatment failure at 24 months | 0 | 1

ADVERSE EVENTS:
Time Frame: Overall study period, up to 24 months
Arm/Group | Aperius™ PercLID™ System | Standalone Decompressive Surgery
Serious Adverse Events (participants affected / at risk) | 26/77 | 25/75
Other Adverse Events (participants affected / at risk) | 53/77 | 57/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aperius™ PercLID™ System (N=77) | Standalone Decompressive Surgery (N=75)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Confusion postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dural tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Neurological and psychiatric procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Facet joint syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculitis lumbosacral (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 6 (6) | 0 (0)
Subdural haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cystocele (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric banding reversal (Surgical and medical procedures) | 0 (0) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 1 (1) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aperius™ PercLID™ System (N=77) | Standalone Decompressive Surgery (N=75)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecal inconsistence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Confusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Dural tear (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Factured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Factured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 8 (8) | 6 (6)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound discence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Biopsy stomach (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (21) | 18 (24)
Buttock pain Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Epicondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Facial bones fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Joint dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (11) | 5 (6)
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Radiculitis lumbosacral (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 4 (4)
Sensory abnormalities NEC (Nervous system disorders) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Impetigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less